CLINICAL TRIAL: NCT03134625
Title: Identification of Metabolite Biomarkers Related to Acute Rejection of Patients With Kidney Transplantation
Brief Title: Metabolite Biomarkers Related to Acute Rejection in Kidney Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1606-069-771
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Kidney Transplantation; Rejection Acute Renal
Keywords: metabolomics; biomarker; acute rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine

SUMMARY:
The development of acute rejection can only be considered in cases with increasing serum creatinine in patients with kidney transplantation. However, the serum creatinine itself is not specific but also accurate for detection of acute rejection. So The specific biomarker is required for acute rejection of kidney transplant. In this study, the investigators will enroll 200 consecutive kidney transplant patients in Seoul National University Hospital and follow up. Serial collection of urine and serum will be done. Acute rejection specific urine metabolite will be found by LC MS/MS.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant patients in Seoul National University Hospital
* Patients with triple maintenance immunosuppression including Tacrolimus, mycophenolate and steroid

Exclusion Criteria:

* History of other organ transplantation
* ABOi and/or crossmatch(+) transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes low or moderate risk kidney transplantation. They should have triple immunosuppression.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-06-28 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
biomarker for acute rejection in kidney transplantation | 1 year
  urine metabolite which is specific for kidney transplant rejection

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea